CLINICAL TRIAL: NCT04230850
Title: The Effects of Stretching Versus Static and Dynamic Cupping on Lumbar Range of Motion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Responsible Party: Principal Investigator, Cathy Arnot, Clinical Associate Professor, University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00092733
Record Dates: First submitted 2019-12-12; First posted 2020-01-18 (Actual); Last update posted 2020-11-16 (Actual); Status verified 2020-11

CONDITIONS: Stiffness; Spine
Keywords: Cupping therapy on lumbar stiffness

STUDY DESIGN:
Intervention Model Description: A parallel design typically compares two or more treatments. Participants are randomly assigned to one of the groups, treatments are administered, and then the results are compared. In this study, individuals will be placed in one of three groups: static stretching group, dynamic cupping group, or stretching group.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The people collecting the data will not be aware of which intervention group the subjects were allocated to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mildly Impaired Group (Active Comparator): This group will consist of participants with 35-50 degrees of lumbar flexion.
  Interventions: Other: Static Cupping; Other: Dynamic Cupping; Other: Stretching
- Moderately Impaired Group (Active Comparator): This group will consist of participants with 20-34 degrees of lumbar flexion.
  Interventions: Other: Static Cupping; Other: Dynamic Cupping; Other: Stretching
- Highly Impaired Group (Active Comparator): This group will consist of participants with less than 20 degrees of lumbar flexion.
  Interventions: Other: Static Cupping; Other: Dynamic Cupping; Other: Stretching

INTERVENTIONS:
Other: Static Cupping — Two cups will be applied unilaterally to the lumbar paraspinals. The skin will be elevated to 1.5 cm ensuring standardized pressure. Cups will remain on the treatment area statically for 4 minutes prior to removal. Another 4 minute bout of identical treatment to the contralateral side will follow. (Participants will be equally dispersed into three treatment groups via stratified randomization).
Other: Dynamic Cupping — One cup will be applied ipsilaterally, raising skin to 1.2 cm of standard pressure. The cup will be continuously moved in a sweeping motion between L1 and L5 within a defined width. This process will be repeated on the other side. Each side will be treated for 4 minutes dynamically for a total treatment duration of 8 minutes. (Participants will be equally dispersed into three treatment groups via stratified randomization).
Other: Stretching — The stretching program performed will involve a double knee to chest stretch, cat stretch, camel stretch, and pelvic tilts. Participants will receive a 30 second rest break between each of the four stretches. (Participants will be equally dispersed into three treatment groups via stratified randomization).

SUMMARY:
The objective of this study is to fill gaps in the literature regarding the effectiveness of cupping therapy on lumbar stiffness. Participants will be recruited from the University of South Carolina and from local clinics in Columbia, South Carolina. Individuals will be classified based on lumbar range of motion limitations, and then they will be equally dispersed into three treatment groups via stratified randomization. These groups include dynamic cupping, static cupping, or stretching. All participants will be assessed prior to selected treatment to obtain baseline values for four measures: back range of motion (BROM), pain pressure threshold (PPT), active straight leg raise (ASLR), and numeric pain rating scale (NPRS). Participants will be given each measure directly after treatment, followed by a follow-up measurement 24 hours after treatment.

DETAILED DESCRIPTION:
Cupping therapy has become recently popular in Western culture due to affordability, lack of invasiveness, and low risk of adverse effects. However, there is insufficient evidence of the effectiveness on this treatment technique on decreasing pain and increasing range of motion. This project aims to help fill the gaps by using a larger sample size and clear methodology.

The aims of the study include to determine if both static and dynamic cupping therapy have a greater effect on BROM, PPT, ASLR, and NRPS as compared to stretching, and if any changes made are maintained to a different degree over a 24 hour period based on treatment. Additional aims of the study include to determine if there is a difference between type of cupping (static vs dynamic) on these four measures. By performing this study, scientific knowledge of cupping therapy will be improved and expanded, thus impacting how it is used in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older, 50 degrees or less of lumbar flexion

Exclusion Criteria:

* Cancer, organ failure, collagen disorders, deep vein thrombosis, pacemakers, bleeding disorders, recent fever

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2020-01-20 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Back Range of Motion | At baseline, immediately following treatment, 24-hour follow up
  The BROM instrument will be used to measure lumbar range of motion in individuals with lumbar stiffness at initial baseline, the change in range of motion immediately following treatment, and any maintained change at 24 hour follow up.

SECONDARY OUTCOMES:
Active Straight Leg Raise | At baseline, immediately following treatment, 24-hour follow up
  The ASLR will be used to assess hamstring flexibility in individuals with lumbar stiffness at initial baseline, the change in hamstring flexibility immediately following treatment, and any maintained change at 24 hour follow up.
Pain Pressure Threshold | At baseline, immediately following treatment, 24-hour follow up
  The Wagner Force Ten FDX Compact Digital Force Gauge hand-held digital algometer will be used to measure pain pressure threshold at initial baseline, the change in pain pressure threshold immediately following treatment, and any maintained change at 24 hour follow up.
Numeric Pain Rating Scale | At baseline, immediately following treatment, 24-hour follow up
  The Numeric Pain Rating Scale will be used to assess pain in individuals with lumbar stiffness at initial baseline, the change in pain immediately following treatment, and any maintained change in 24 hour follow up. Individuals will be asked to rate their current pain level on a scale of 0-10, with "0" representing no pain and "10" representing the worst pain imaginable.

CONTACTS AND LOCATIONS:
Overall Officials: Cathy Arnot, DPT, Principal Investigator — University of South Carolina
Locations (1):
- University of South Carolina, Columbia, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No
All data collected will be analyzed and interpreted only by the investigators listed for University of South Carolina.

REFERENCES:
- [Background] Rozenfeld E, Kalichman L. New is the well-forgotten old: The use of dry cupping in musculoskeletal medicine. J Bodyw Mov Ther. 2016 Jan;20(1):173-178. doi: 10.1016/j.jbmt.2015.11.009. Epub 2015 Dec 1. PMID 26891653
- [Background] Markowski A, Sanford S, Pikowski J, Fauvell D, Cimino D, Caplan S. A pilot study analyzing the effects of Chinese cupping as an adjunct treatment for patients with subacute low back pain on relieving pain, improving range of motion, and improving function. J Altern Complement Med. 2014 Feb;20(2):113-7. doi: 10.1089/acm.2012.0769. Epub 2013 Dec 3. PMID 24299469
- [Background] Shum GL, Crosbie J, Lee RY. Symptomatic and asymptomatic movement coordination of the lumbar spine and hip during an everyday activity. Spine (Phila Pa 1976). 2005 Dec 1;30(23):E697-702. doi: 10.1097/01.brs.0000188255.10759.7a. PMID 16319739
- [Background] Coyle PC, Velasco T, Sions JM, Hicks GE. Lumbar Mobility and Performance-Based Function: An Investigation in Older Adults with and without Chronic Low Back Pain. Pain Med. 2017 Jan 1;18(1):161-168. doi: 10.1093/pm/pnw136. PMID 27346888
- [Background] Clarkson, H. M. (2013). Musculoskeletal assessment: Joint motion and muscle testing (3rd ed.). Philadelphia: Wolters Kluwer & Lippincot Williams & Wilkins.
- [Background] Kuo YL, Tully EA, Galea MP. Kinematics of sagittal spine and lower limb movement in healthy older adults during sit-to-stand from two seat heights. Spine (Phila Pa 1976). 2010 Jan 1;35(1):E1-7. doi: 10.1097/BRS.0b013e3181c47a0e. PMID 20042941
- [Background] Meucci RD, Fassa AG, Faria NM. Prevalence of chronic low back pain: systematic review. Rev Saude Publica. 2015;49:1. doi: 10.1590/S0034-8910.2015049005874. Epub 2015 Oct 20. PMID 26487293
- [Background] Yang H, Haldeman S, Lu ML, Baker D. Low Back Pain Prevalence and Related Workplace Psychosocial Risk Factors: A Study Using Data From the 2010 National Health Interview Survey. J Manipulative Physiol Ther. 2016 Sep;39(7):459-472. doi: 10.1016/j.jmpt.2016.07.004. Epub 2016 Aug 25. PMID 27568831
- [Background] Thiese MS, Hegmann KT, Wood EM, Garg A, Moore JS, Kapellusch JM, Foster J, Greene T, Stoddard G, Biggs J; BackWords Study Team. Low-back pain ratings for lifetime, 1-month period, and point prevalences in a large occupational population. Hum Factors. 2014 Feb;56(1):86-97. doi: 10.1177/0018720813493641. PMID 24669545
- [Background] Luckhaupt SE, Dahlhamer JM, Gonzales GT, Lu ML, Groenewold M, Sweeney MH, Ward BW. Prevalence, Recognition of Work-Relatedness, and Effect on Work of Low Back Pain Among U.S. Workers. Ann Intern Med. 2019 Aug 20;171(4):301-304. doi: 10.7326/M18-3602. Epub 2019 May 14. PMID 31083729
- [Background] Hartvigsen J, Hancock MJ, Kongsted A, Louw Q, Ferreira ML, Genevay S, Hoy D, Karppinen J, Pransky G, Sieper J, Smeets RJ, Underwood M; Lancet Low Back Pain Series Working Group. What low back pain is and why we need to pay attention. Lancet. 2018 Jun 9;391(10137):2356-2367. doi: 10.1016/S0140-6736(18)30480-X. Epub 2018 Mar 21. PMID 29573870
- [Background] Delitto A, George SZ, Van Dillen L, Whitman JM, Sowa G, Shekelle P, Denninger TR, Godges JJ; Orthopaedic Section of the American Physical Therapy Association. Low back pain. J Orthop Sports Phys Ther. 2012 Apr;42(4):A1-57. doi: 10.2519/jospt.2012.42.4.A1. Epub 2012 Mar 30. PMID 22466247
- [Background] Kisner, C., Colby, L. A., & Borstad, J. (2017). Therapeutic exercise: Foundations and techniques. Fa Davis.
- [Background] Nelson RT, Bandy WD. Eccentric Training and Static Stretching Improve Hamstring Flexibility of High School Males. J Athl Train. 2004 Sep;39(3):254-258. PMID 15496995
- [Background] Page P. Current concepts in muscle stretching for exercise and rehabilitation. Int J Sports Phys Ther. 2012 Feb;7(1):109-19. PMID 22319684
- [Background] Bandy WD, Irion JM, Briggler M. The effect of time and frequency of static stretching on flexibility of the hamstring muscles. Phys Ther. 1997 Oct;77(10):1090-6. doi: 10.1093/ptj/77.10.1090. PMID 9327823
- [Background] Roussel NA, Nijs J, Truijen S, Smeuninx L, Stassijns G. Low back pain: clinimetric properties of the Trendelenburg test, active straight leg raise test, and breathing pattern during active straight leg raising. J Manipulative Physiol Ther. 2007 May;30(4):270-8. doi: 10.1016/j.jmpt.2007.03.001. PMID 17509436
- [Background] Breum J, Wiberg J, Bolton JE. Reliability and concurrent validity of the BROM II for measuring lumbar mobility. J Manipulative Physiol Ther. 1995 Oct;18(8):497-502. PMID 8583171
- [Background] Phattharasupharerk, S., Purepong, N., & Siriphorn, A. Inter-and Intra-Rater Reliability of the Back Range of Motion Instrument (BROM II) for Measuring Lumbar Mobility in Persons with Sedentary Lifestyle.
- [Background] Fischer AA. Pressure algometry over normal muscles. Standard values, validity and reproducibility of pressure threshold. Pain. 1987 Jul;30(1):115-126. doi: 10.1016/0304-3959(87)90089-3. PMID 3614975
- [Background] Potter, L., McCarthy. C., Oldham, J. Algometer reliability in measuring pain thresholds over normal spinal muscles to allow quantification of anti-nociceptive treatment effects. International Journal of Osteopathic Medicine, 9 (2006), pp. 113-119.
- [Background] Nussbaum EL, Downes L. Reliability of clinical pressure-pain algometric measurements obtained on consecutive days. Phys Ther. 1998 Feb;78(2):160-9. doi: 10.1093/ptj/78.2.160. PMID 9474108
- [Background] Liebenson C, Karpowicz AM, Brown SH, Howarth SJ, McGill SM. The active straight leg raise test and lumbar spine stability. PM R. 2009 Jun;1(6):530-5. doi: 10.1016/j.pmrj.2009.03.007. PMID 19627942
- [Background] Gajdosik RL, LeVeau BF, Bohannon RW. Effects of ankle dorsiflexion on active and passive unilateral straight leg raising. Phys Ther. 1985 Oct;65(10):1478-82. doi: 10.1093/ptj/65.10.1478. PMID 4048283
- [Background] Childs JD, Piva SR, Fritz JM. Responsiveness of the numeric pain rating scale in patients with low back pain. Spine (Phila Pa 1976). 2005 Jun 1;30(11):1331-4. doi: 10.1097/01.brs.0000164099.92112.29. PMID 15928561
- [Background] Chen HM, Wang HH, Chen CH, Hu HM. Effectiveness of a stretching exercise program on low back pain and exercise self-efficacy among nurses in Taiwan: a randomized clinical trial. Pain Manag Nurs. 2014 Mar;15(1):283-91. doi: 10.1016/j.pmn.2012.10.003. Epub 2012 Dec 23. PMID 23266331